CLINICAL TRIAL: NCT02701010
Title: Comparative Effectiveness of Three Different Teaching Methods in Behavioural Therapy Program for Female Overactive Bladder: A Randomized Controlled Trial
Brief Title: Behavioural Therapy Program for Female Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Sercan YILMAZ, Medical Doctor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: -1491-160-12/1648.4-5263
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Urinary Bladder, Overactive
Keywords: behavioral therapy; overactive bladder; urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Active Comparator): Structured training and leaflet
  Interventions: Behavioral: Structured training and leaflet
- Group 2 (Active Comparator): Structured training
  Interventions: Behavioral: Structured training
- Group 3 (Active Comparator): Leaflet
  Interventions: Behavioral: Leaflet
- Group 4 (Sham Comparator): Control group
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Structured training and leaflet — The patients who were given both "explanatory verbal instructions of the educational leaflet on the structured behavioural therapy for iOAB" by continence nurse and the educational leaflet were included in this group.
  Arms: Group 1
Behavioral: Structured training — The patients who were given only "explanatory verbal instructions of the educational leaflet on the structured behavioural therapy" by continence nurse were included in this group.
  Arms: Group 2
Behavioral: Leaflet — The patients who were given "only educational leaflet" were included in this group.
  Arms: Group 3
Behavioral: Control Group — Patients who were given unstructured explanations about continence care by a healthcare worker were included in control group.
  Arms: Group 4

SUMMARY:
Researchers aimed to identify the effectiveness of three methods of patient education for behavioral therapy (BT), including verbal instructions combined with a leaflet on a structured training program of BT, only verbal instructions on a structured training and only a leaflet on a structured BT training. Therefore, a randomized controlled trial was designed to compare effectiveness of those methods of patient education in BT based on the two validated patient- reported outcome measures (PROMs) for women with overactive bladder.

Idiopathic overactive bladder (iOAB) symptoms in female patients are perceived as normal, which does not threaten life and not require to be treated immediately. It is necessary to raise the awareness of iOAB on women. The education and consultancy role of continence nurses is important in the treatment and care of urinary incontinence (UI) associated with iOAB. In the study, it was seen that the training to be provided to patients is helpful regardless of the teaching method used. Also it was found that the method of verbal instructions in the form of a structured training plus giving a leaflet to patient is the most effective method of BT for female iOAB.

DETAILED DESCRIPTION:
Behavioural therapy (BT) is the first-line treatment for urinary incontinence including idiopathic overactive bladder (iOAB) syndrome. It requires education of the actively participated patient as well as time and effort from the clinician. However, the most effective method for patient education in BT remains unclear. Researchers designed a randomized controlled trial to compare effectiveness of 3 different methods of patient education in BT for women with overactive bladder.

The sample of the study consisted of 60 iOAB female patients who applied to urogynecology clinic between November 2012 and April 2013. These patients were equally randomized into 4 groups of teaching models for BT. Group I included the patients educated by a continence nurse's verbal instructions in the form of a structured training including bladder training, bladder control strategies, pelvic floor muscle training and lifestyle changes and a leaflet containing information stated in structured training, group II included the patients taught by a continence nurse as the only verbal structured training, group III included the patients who were given only the leaflet and group IV was the control group consisted of female iOAB patients who were given an unstructured training by a healthcare worker with no specific experience in continence care.

ELIGIBILITY:
Eligible participants were all ambulatory adults aged 18 or over with predominant iOAB syndrome with or without stress urinary incontinence (the number of urgency and urgency incontinence episodes exceeded the number of stress incontinence episodes and other accidents in bladder diary), who were candidates for behavioural therapy as a first-line treatment after initial clinical assessment, including history, physical examination, symptom questionnaires, 3-day bladder diary, repeated uroflowmetry and postvoid residual measurements for all patients and urodynamics for some patients with a suspicion of presence of the exclusion criteria.

Exclusion criteria were pregnancy, suspected neurogenic disease, stress predominant mixed urinary incontinence, continuous urinary leakage, previous anti-incontinence surgery, voiding dysfunction (PVR> 100 ml), genitourinary malignancies, current or previous behavioural therapy programs, previous or current use of antimuscarinic agents, symptomatic pelvic organ prolapse, severe co-morbidities such as congestive heart failure, chronic renal failure, impaired cognitive functions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Urogenital Distress Inventory (UDI-6) | baseline to 6 or 8 weeks
  improvement in bladder functions at 6-8 weeks of the intervention compared to baseline
Incontinence Impact Questionnaire (IIQ-7) | baseline to 6 or 8 weeks
  improvement in bladder functions at 6-8 weeks of the intervention compared to baseline

SECONDARY OUTCOMES:
Urinary Incontinence-Specific Quality of Life Instrument (I-QOL) | baseline to 6 or 8 weeks
  positive changes in quality of life at 6-8 weeks of the intervention compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Military Medical Academy, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] Sacco E, Tienforti D, D'Addessi A, Pinto F, Racioppi M, Totaro A, D'Agostino D, Marangi F, Bassi P. Social, economic, and health utility considerations in the treatment of overactive bladder. Open Access J Urol. 2010 Feb 11;2:11-24. doi: 10.2147/rru.s4166. PMID 24198609
- [Background] Abrams P. CL, Khoury S, Wein A, ed Incontinence 4th Edition. 21 ed. Paris: Health Publication; 2009. 4th International Consultation on Incontinence.
- [Background] Cam C, Sakalli M, Ay P, Cam M, Karateke A. Validation of the short forms of the incontinence impact questionnaire (IIQ-7) and the urogenital distress inventory (UDI-6) in a Turkish population. Neurourol Urodyn. 2007;26(1):129-33. doi: 10.1002/nau.20292. PMID 17083117
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Patrick DL, Martin ML, Bushnell DM, Yalcin I, Wagner TH, Buesching DP. Quality of life of women with urinary incontinence: further development of the incontinence quality of life instrument (I-QOL). Urology. 1999 Jan;53(1):71-6. doi: 10.1016/s0090-4295(98)00454-3. PMID 9886591
- [Background] Ozerdogan N, Beji NK, Yalcin O. Urinary incontinence: its prevalence, risk factors and effects on the quality of life of women living in a region of Turkey. Gynecol Obstet Invest. 2004;58(3):145-50. doi: 10.1159/000079422. Epub 2004 Jun 29. PMID 15237249
- [Background] Available from: https://www.sealedenvelope.com/simple-randomiser/v1/lists, available date: 01.11.2012
- [Background] Subak LL, Goode PS, Brubaker L, Kusek JW, Schembri M, Lukacz ES, Kraus SR, Chai TC, Norton P, Tennstedt SL; Urinary Incontinence Treatment Network. Urinary incontinence management costs are reduced following Burch or sling surgery for stress incontinence. Am J Obstet Gynecol. 2014 Aug;211(2):171.e1-7. doi: 10.1016/j.ajog.2014.03.012. Epub 2014 Mar 11. PMID 24631433
- [Background] Lucas MG, Bosch RJ, Burkhard FC, Cruz F, Madden TB, Nambiar AK, Neisius A, de Ridder DJ, Tubaro A, Turner WH, Pickard RS; European Association of Urology. EAU guidelines on assessment and nonsurgical management of urinary incontinence. Eur Urol. 2012 Dec;62(6):1130-42. doi: 10.1016/j.eururo.2012.08.047. Epub 2012 Aug 31. PMID 22985745
- [Background] Botlero R, Urquhart DM, Davis SR, Bell RJ. Prevalence and incidence of urinary incontinence in women: review of the literature and investigation of methodological issues. Int J Urol. 2008 Mar;15(3):230-4. doi: 10.1111/j.1442-2042.2007.01976.x. PMID 18304218
- [Background] Elbiss HM, Osman N, Hammad FT. Social impact and healthcare-seeking behavior among women with urinary incontinence in the United Arab Emirates. Int J Gynaecol Obstet. 2013 Aug;122(2):136-9. doi: 10.1016/j.ijgo.2013.03.023. Epub 2013 Jun 10. PMID 23764126
- [Background] Tsai YC, Liu CH. Urinary incontinence among Taiwanese women: an outpatient study of prevalence, comorbidity, risk factors, and quality of life. Int Urol Nephrol. 2009 Dec;41(4):795-803. doi: 10.1007/s11255-009-9523-3. Epub 2009 Feb 6. PMID 19199071
- [Background] Hsieh CH, Su TH, Chang ST, Lin SH, Lee MC, Lee MY. Prevalence of and attitude toward urinary incontinence in postmenopausal women. Int J Gynaecol Obstet. 2008 Feb;100(2):171-4. doi: 10.1016/j.ijgo.2007.08.013. Epub 2007 Oct 31. PMID 17977542
- [Background] Hunskaar S. A systematic review of overweight and obesity as risk factors and targets for clinical intervention for urinary incontinence in women. Neurourol Urodyn. 2008;27(8):749-57. doi: 10.1002/nau.20635. PMID 18951445
- [Background] Hagglund D, Walker-Engstrom ML, Larsson G, Leppert J. Reasons why women with long-term urinary incontinence do not seek professional help: a cross-sectional population-based cohort study. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Nov;14(5):296-304; discussion 304. doi: 10.1007/s00192-003-1077-9. Epub 2003 Aug 29. PMID 14618304
- [Background] O'Donnell M, Lose G, Sykes D, Voss S, Hunskaar S. Help-seeking behaviour and associated factors among women with urinary incontinence in France, Germany, Spain and the United Kingdom. Eur Urol. 2005 Mar;47(3):385-92; discussion 392. doi: 10.1016/j.eururo.2004.09.014. Epub 2004 Nov 21. PMID 15716205
- [Background] Subak LL, Quesenberry CP, Posner SF, Cattolica E, Soghikian K. The effect of behavioral therapy on urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2002 Jul;100(1):72-8. doi: 10.1016/s0029-7844(02)01993-2. PMID 12100806
- [Background] Kök G, Şenel N, Akyüz A. Nurses' roles in identifying urinary incontinence and its effects on social life. Int J Urol Nurs 2008;2:119-124.
- [Background] Altaweel W, Alharbi M. Urinary incontinence: prevalence, risk factors, and impact on health related quality of life in Saudi women. Neurourol Urodyn. 2012 Jun;31(5):642-5. doi: 10.1002/nau.22201. Epub 2012 Mar 13. PMID 22415626
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598